CLINICAL TRIAL: NCT03511235
Title: Clinical Outcomes in Men With Prostate Cancer Who Selected Active Surveillance Using Prolaris® Testing
Acronym: URO-009Low
Status: Completed | Type: Observational
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: URO-009
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medicare is requesting outcome data on patients who received Prolaris testing and were prescribed active surveillance (AS). In order to ensure appropriate patient care, it is important to understand how this added prognostic information influences the selection and durability of AS and corresponding clinical outcomes. To address this knowledge gap, this study will evaluate how frequently men with low disease-specific mortality (DSM) risk based on Prolaris CCR score and who meet NCCN low-risk criteria initially select AS (AS selection). This study also will assess how long Prolaris-tested men who initially select AS remain on this course before proceeding to definitive treatment (AS durability), and whether AS duration impacts biochemical recurrence (BCR) and metastasis risk in these men. This retrospective, observational and multi-site study will combine patient CCR scores with longitudinal clinical data to address these questions.

DETAILED DESCRIPTION:
This is a multicenter, retrospective, observational study in men diagnosed with localized PrCa who had Prolaris testing prior to the treatment decision. The study will collect demographic, clinical, pathologic, and Prolaris test data from medical records and Myriad's Prolaris database.

The primary objective of this study is to evaluate the rate of BCR or metastasis, whichever occurs first, among Prolaris-tested men who were at low risk of DSM (≤3.2%), who also met NCCN low-risk criteria, and who were initially treated with AS.

The secondary objectives of the study are to evaluate the frequency of AS selection among all men who had low DSM risk, as determined by Prolaris testing and AS durability among Prolaris-tested men with low DSM risk who selected and initiated this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with localized PrCa at participating sites between January 1, 2013 and August 1, 2017.
* Have undergone Prolaris testing and have a CCR score with estimated DSM risk ≤3.2%.
* Have NCCN low-risk disease2.

Exclusion Criteria:

* Received any therapy other than 5α-reductase inhibitor (5-ARI) prior to diagnostic biopsy.
* Over 80 years of age at diagnosis.
* History of hypogonadism at the time of diagnosis.
* Co-occurring malignancy, excluding non-melanoma skin cancer.
* Enrolled in another investigational study.

Max Age: 80 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Not based on self-representation of gender identity
Study Population: Prolaris-tested men diagnosed with low-risk prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of BCR or metastasis after selection of active surveillance (AS) | Up to five years post Prolaris report
  This study will evaluate how frequently men with low disease-specific mortality (DSM) risk based on Prolaris CCR score and who meet NCCN low-risk criteria initially select AS (AS selection). This study also will assess how long Prolaris-tested men who initially select AS remain on this course before proceeding to definitive treatment (AS durability), and whether AS duration impacts biochemical recurrence (BCR) and metastasis risk in these men.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan M Dechairo, PhD, Study Director — Myriad Genetics, Inc.
Locations (8):
- United States (8):
  - Arkansas Urology, Little Rock, Arkansas
  - Pacific Urology, Concord, California
  - Kar Urology, Orange, California
  - Golden Gate Urology, San Francisco, California
  - Urological Associates, Colorado Springs, Colorado
  - University of Michigan Urology Cancer Center, Ann Arbor, Michigan
  - Dr. Jeffrey Glaser, Urologist, Lake Saint Louis, Missouri
  - Memorial Sloane Kettering Cancer Center, New York, New York